CLINICAL TRIAL: NCT00338702
Title: A Randomized, Controlled Trial of Autologous Platelet Gel Treatment in Diabetic Foot Ulcers
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Industry support and funding not forthcoming
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1_James L Mahoney
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2015-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic; Foot; Ulcer; Autologous; Platelet; Gel
MeSH Terms: conditions — Diabetic Foot; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Autologous Platelet Gel

SUMMARY:
Foot ulcers represent a significant common complication in patients with diabetes. Wound healing is a challenge. Some wounds do not respond to the best practices in wound care. Considerable effort has been directed at therapies to improve the rate of healing.

There are a variety of growth factors which have been used to stimulate wound healing. Human platelets are an autologous source of growth factors which probably can stimulate healing. Autologous platelet gel (APG) is prepared by centrifugation of autologous human whole blood. APG is rich in platelet growth factors. This study will investigate the potential improvement in wound healing with this material in diabetic foot ulcers.

This study will compare the use of autologous platelet gel ( study group) and standard care ( control group) in the treatment of diabetic plantar forefoot ulcers. This study will also compare the cost and quality of life in the two groups.

Objectives of the study:

* To determine if topical APG (autologous platelet gel) is beneficial in the treatment of diabetic foot ulcers.
* To determine if it will result in a faster rate of wound healing.
* To determine if it will improve the quality of life in patients with diabetic foot ulcers.

DETAILED DESCRIPTION:
Study Design This will be a single center, randomized, controlled, prospective study comparing the use of autologous platelet gel (study group) and traditional moist dressing (control group) in the treatment of plantar forefoot ulcers.

Specific Aims Primary - Facilitation of healing of diabetic foot ulcers Secondary - Reduction in amputations and average total cost of care. Determine the impact of diabetic ulcers on patients' quality of life Research Background Foot ulcers represent a significant common complication in patients with diabetes. It is estimated that twenty percent of all patients with diabetes develop a foot ulcer which may subsequently lead to below knee amputation. 85 % of them preceded by non-healing foot ulcers.

Health care costs associated with diabetic foot wound management are staggering. Armstrong et al (1998) reported that wound care for foot ulcer patients over a two year period had mean cost of $27,000.00 U.S. In Toronto, the average cost of below knee amputations, including hospitalization and rehabilitation, is $40,000.00.

Wound healing in the context of diabetes is a challenge for both the health care provider and the patient. In a systematic review conducted by Margolis et al (1999), wound healing outcomes using best practices have yielded only 24% at 12 weeks, 31% in 20 weeks.

Falanga & Sabolinski (2001) identified that initial wound size reduction of 0.1 cm/week is highly predictive of wound closure whereas initial healing rates 0.06 cm or less predict non-healing. Similarly, 51% percent reduction in 4 weeks was found to be a good predictor of achieving wound closure (Margolis et al, 1999). Some wounds do not respond and considerable effort has been directed at therapies to improve the rate of healing in this situation.

A variety of growth factors which have been used to stimulate wound healing. Human platelets are an autologous source which probably can stimulate healing. Autologous platelet gel (APG) is a material presently utilized as a tissue adhesive. It is derived from platelet rich plasma (PRP) that was first developed in the early 1990's to primarily address acute surgical hemostatic and wound healing problems.

APG is prepared by centrifugation of autologous human whole blood, which initially separates it into three components: packed red cells, platelet poor plasma, and platelet rich plasma (PRP). PRP has two to eight times the normal concentration of platelets in human blood. The key element that differentiates APG from traditional fibrin glue is the presence of concentrated platelets rich in platelet growth factors. These important elements of the blood, in an increased concentration are potentially helpful in improving the rate of wound healing. This study will investigate the potential improvement in wound healing with APG in diabetic foot ulcers.

Rationale for the Research

* To determine if topical APG (autologous platelet gel) is beneficial in the treatment of diabetic foot ulcers.
* To determine if it will result in a faster rate of wound healing.
* To determine if it will improve the quality of life in patients with diabetic foot ulcers Study Population Subjects for this study will be recruited from our patient population. Fifty patients will be randomized to one of the two treatment groups 9 study and control).

Inclusion Criteria

1. >18 years of age
2. Type I or Type II Diabetes
3. Plantar forefoot ulcer(s) beneath metatarsal head or toe ulcer which has been present for at least 4 weeks, and has received best practice care
4. Evidence of adequate arterial perfusion: Toe plethysmography reading of ≥ 45 mmHg or Transcutaneous oxygen measurement of ≥ 30mmHg
5. Patient is appropriately offloaded (contact cast, pneumatic walking cast)
6. Infection and/or osteomyelitis have been ruled out or are being treated
7. Platelet count greater than150,000/mm3
8. Orthopedic assessment has been completed to rule out mechanical source of ulceration
9. Patients with following skeletal deformities could be included -

   1. Tendoachillis contracture - after tendoachillis contracture lengthening has been done
   2. Charcot arthropathy with concurrent surgical intervention
   3. Toe deformities ( hallus valgus, significant claw toe deformities) with/after surgical intervention
   4. Major axial malalignment (hindfoot varus/valgas, pes planus, pes cavus) with/after surgical intervention
10. Patients taking clopidogrel (Plavix) and aspirin could be included in the study. Patients taking aspirin for non medical reason will be asked to discontinue the medicine one week before the start of treatment.

Exclusion Criteria

1. TcPO2 <30 mmHg and/or toe plethysmography readings of less than 45 mmHg
2. Limb ischemia requiring re-vascularization or impending amputation
3. Untreated wound infection or osteomyelitis
4. Bleeding disorders, hemophilia, sickle cell disease, thrombocytopenia, and leukemia or blood dyscrasias
5. Anemia with hemoglobin level less than 100 g/L will be included as exclusion criteria.
6. Patient is taking immunosuppressive agents (e.g. corticosteroids, chemotherapeutic agents, transplant medications)
7. Current treatment for malignancy or neoplastic disease or collagen vascular disease
8. Patients taking anticoagulants like heparin or coumadin or others which may hinder in clot (thrombin) formation
9. Patient has a highly communicable disease or diseases that may limit follow - up (e.g. immuno-compromised conditions, hepatitis, active tuberculosis)
10. Ulcers resulting from electrical, chemical, radiation burns
11. Serum creatinine level >110 umol/L
12. HbA1c > 9%
13. Currently participating in another investigation study
14. Ulcer with exposed bone or tendon Withdrawal Criteria

1. The patient may be withdrawn from the study at the discretion of the investigator if judged noncompliant with study procedures or worsening patient condition 2. Detection of osteomyelitis that is not treatable by debridement and antibiotics at the discretion of the investigator 3. Development of progressive wound necrosis Experimental Methods For study purposes, diabetic foot ulcer will be a wound on the plantar aspect of the foot which has not responded to at least 4 weeks of best practice care. Complete wound closure will be defined as skin closure (100% re-epithelization) without drainage or dressing requirements.

Patients seeking treatment for diabetic foot ulcers that meet the entry criteria will be considered for the study. Patients will be randomized to either the STUDY or the CONTROL group with a 1:1 control to study ratio.

STUDY Group Patients will have APG (autologous platelet gel) applied to the wound in accordance with institutional treatment protocols and manufacturer's guidelines. Dressing changes will occur at least three times a week.

Method of preparing and application of autologous platelet gel is as follows -

1. Obtain 54 cc of whole blood into a 60 cc syringe with 6 cc of citrate anticoagulant through standard blood draw technique.
2. Slowly load blood filled syringe into GPS II unit's centre port. And centrifuge for 15 minutes.
3. Draw PRP (Platelet Rich Plasma) concentrate from GPS II unit into a 10 cc syringe.
4. Prepare the wound bed through sharp excision of the eperbole, necrotic tissue & wound bed.
5. Aspirate PPP (Platelet Poor Plasma) from GPSII unit in to a 30 ml syringe.
6. Inject Thrombin Reagent (5 cc of CaCl2) to Thrombin Processing Device and then add 11 cc of the PPP from the syringe and after mixing let it stand for 20 minutes.
7. Draw 1 cc of thrombin/CaCl2 solution into a 1 cc syringe from Thrombin Processing Device.
8. Connect syringe with PRP and syringe with thrombin/CaCl2 to a dual sprayer
9. Spray solutions over entire wound bed. Protect surrounding skin (but not into the wound) with barrier film.
10. Apply a semi-permeable, film-type dressing as primary dressing. Leave dressing in place for 3-7 days.
11. The affected limb will receive offloading in the form of a total contact cast, a pneumatic walking cast or wheelchair.
12. After the first dressing with APG the wound will be dressed with a moist dressing, similar to control group dressings. The dressings will be changed daily or on a Monday-Wednesday-Friday routine based on the level of exudates.

CONTROL Group

Weekly standard therapy alone as follows:

1. Any debridement deemed necessary is performed
2. Ulcer-site will be dressed with a moist dressing such as cadexamer iodine ointment (Iodosorb) and an absorbent covering dressing that is moisture retentive. Acceptable other control group dressing types are: alginates, hydrogels and hydrocolloids and saline gauze. The dressing will be changed daily or on a Monday-Wednesday-Friday routine based on the level of exudate.
3. The affected limb will receive offloading in the form of a total contact cast, a pneumatic walking cast or wheelchair.

Treatment Phase of the Study: Treatment in both groups will continue until the wound is successfully closed.

At 12 weeks (3 months) wounds from both control and treatment groups will be evaluated. If the wound does not show any signs of improvement (wound closure by 50% at 3 months) the wound will be considered as a treatment failure and it will be treated with alternate dressing according to hospital standard of care. These wounds will be followed every month till they close.

6-Month and 12 month follow-up: For patients who achieved wound closure at 12 weeks, or later the wound site will undergo an examination for recurrence.

No patient will remain in the study for longer than 12 months (total study duration).

Clinical Assessments A. Wound Debridement All wounds under study will be surgically debrided The wound may be debrided by autolysis or sharp wound debridement as tolerated.

B. Laboratory Testing Up to seven days prior to the initiation of protocol treatment, blood samples will be taken to determine serum pre-albumin, albumin and creatinine levels. If the pre-albumin is <16 mg/dl (<160 mg/L) or the albumin level is <3 g/dl (<30 g/L), nutritional supplementation will be started. The tests will be repeated at 12 weeks or at the time of wound closure which ever comes first. Determination of HbA1c will be performed up to 30 days prior to initiation of protocol treatment, and at 12 weeks or at the time of wound closure which ever comes first.

Bacterial culture will be done at Day 0. Additional cultures may be obtained as clinically indicated.

C. Wound Examination Ulcers will be examined at Days 0, 7 (1 wk), 14 (2wk), 28 (4wk) , 56 (8wk), 84 (12wk), 6 and 12 month follow up visits.

The ulcer will be classified using the University of Texas Scale Diabetic Foot ulcer Classification System.

The ulcer will be evaluated using following criteria:

* Time to closure
* Granulation tissue formation will be categorically estimated in percentages and recorded as 0-10%, 11-25 %, 26-50 %, 51-75 % or 75-100%
* Eschar and necrotic tissue estimation
* Wound edge evaluation - evidence of epithelial tissue
* Amount ( scant, moderate, copious) and quality ( serous, purulent, sanguinous) of wound exudate
* Evidence of infection ( erythema, odor, pain at ulcer site, ulcer deterioration)
* Wound assessment will be done, to include measurement of standard wound width, length and depth. Wound tracings will be performed using the Visitrak and depth will be measured by the placement of a wooden end of sterile cotton tipped applicator into the deepest part of the wound, withdrawing and measuring that length
* Ulcer photographs will be taken using a digital camera. D. Wound Pain Assessments - The patient will complete the wound pain assessment using a visual analog scale (VAS) at all study visits. The pain assessment will be done prior to and within one-half hour after the wound dressing changes. Pain medication use will be documented.

E. Documentation of Dressings - The number and type of dressings used will be documented by the health care professional taking care of the patient.

F. Cost - Frequency of dressing changes and estimates of material cost and nursing time will be documented Data Collection/Study Visit Procedures Visit 1 (Day -7 to Day 0) Screening Patients will be screened and data will be collected for demographic details, relevant medical and surgical history, lab values, results of vascular studies and Plastic and / or Orthopedic Surgeons' consultations Visit 2 (Day 0) Randomization/Treatment It will take place within 7 days after Visit 1. Patients will be randomized. Wounds will be assessed, photographed and measured and data will be collected.

Visit 3, 4, 5, 6, and 7 (week 1 (05 days), week 2, 4, 8 and 12) Wounds will be assessed, photographed and measured and data will be collected. Number of dressing changes per week, materials used and the occupation of person performing the dressing change will be documented. The time to definitive wound closure will be recorded. Pre-albumin, albumin creatinine and HbA1c will be tested at week 12. Ulcer recurrence and its cause will be documented.

Visit 8 and 9 (6 Month and12 Month Follow-up) Assessment of Recurrence These visits will occur at 6 months and 12 months for both treatment groups. The wound will be examined for recurrence or determination of wound status. Information about patient's quality of life using Cardiff Wound Impact questionnaire, 6 months after healing of the ulcer will be collected.

Adverse Events Through out the study period adverse events, also termed "study events" and "adverse experiences" and serious adverse events will be recorded.

Statistical Analysis Endpoints will include: time to 25% percent closure at 6 weeks, time to 50% closure at 12 weeks and time to definitive closure Analyses will include - time to 50-percent-closure, time to definitive closure, percentage of wounds closed at study calendar time points/visits, number of dressing changes and impact of diabetic foot ulcer on the quality of life Survival analysis, ANOVA/ANCOVA, and non-parametric analysis will be used. A repetitive measurement analysis will also be applied. Ordinal Categorical Analysis will be performed on data from Cardiff Wound Impact Schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patient is greater than 18 years of age
* Patient has Type I or Type II Diabetes
* Patient must be able to understand English (self or translator) and give written, informed consent
* Patient has a plantar forefoot ulcer(s) beneath metatarsal head or toe ulcer which has been present for at least 4 weeks, and has received best practice care
* Evidence of adequate arterial perfusion: Toe plethysmography reading of

  * 45 mmHg or Transcutaneous oxygen measurement of ≥ 30mmHg
* Patient is appropriately offloaded (contact cast, pneumatic walking cast)
* Infection and/or osteomyelitis have been ruled out or are being treated
* Patients must have a platelet count greater than150,000/mm3
* Orthopedic assessment has been completed to rule out mechanical source of ulceration
* Patients with following skeletal deformities could be included -

  1. Tendoachillis contracture - after tendoachillis contracture lengthening has been done
  2. Charcot arthropathy with concurrent surgical intervention
  3. Toe deformities ( hallus valgus, significant claw toe deformities) with/after surgical intervention
  4. Major axial malalignment (hindfoot varus/valgas, pes planus, pes cavus) with/after surgical intervention
* Patients taking clopidogrel (Plavix) and aspirin could be included in the study. Patients taking aspirin for non medical reason will be asked to discontinue the medicine one week before the start of treatment.

Exclusion Criteria:

* TcPO2 <30 mmHg and/or toe plethysmography readings of less then 45 mmHg
* Limb ischemia requiring re-vascularization or impending amputation
* Untreated wound infection or osteomyelitis
* Bleeding disorders, hemophilia, sickle cell disease, thrombocytopenia,and leukemia or blood dyscrasias
* Anemia with hemoglobin level less than 100 g/L will be included as exclusion criteria.
* Patient is taking immunosuppressive agents (e.g. corticosteroids, chemotherapeutic agents, transplant medications)
* Current treatment for malignancy or neoplastic disease or collagen vascular disease
* Patient has a highly communicable disease or diseases that may limit follow - up (e.g. immuno-compromised conditions, hepatitis, active tuberculosis)
* Patients taking anticoagulants like heparin or coumadin or others which may hinder in clot (thrombin) formation
* Ulcers resulting from electrical, chemical, radiation burns
* Serum creatinine level >110 umol/L
* HbA1c > 9%
* Currently participating in another investigation study
* Ulcer with exposed bone or tendon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Time to 25% percent closure at 6 weeks
Time to 50% closure at 12 weeks
Time to definitive closure

CONTACTS AND LOCATIONS:
Overall Officials: James L Mahoney, MD, FRCSC, Principal Investigator — Unity Health Toronto; Timothy R Daniels, MD, FRCSC, Principal Investigator — St. Michael Hospital
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada